CLINICAL TRIAL: NCT07280468
Title: Endotype DIrected Treatment for OSA in Down Syndrome
Acronym: EDIT OSA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Daniel A. Combs, Associate Professor of Pediatrics and Medicine, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00007297; IDD-2024C1-37111 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2025-11-23; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea (OSA); Down Syndrome
Keywords: Down syndrome; obstructive sleep apnea; ato-oxy; precision medicine; oxygen; atomoxetine; oxybutynin
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome | interventions — Atomoxetine Hydrochloride; oxybutynin; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uniform therapy (ato-oxy) (Active Comparator): All participants receive the combination of atomoxetine and oxybutynin (ato-oxy) once nightly
  Interventions: Drug: ato-oxy
- Endotype Directed Treatment (Experimental): Participants receive either atomoxetine and oxybutynin (ato-oxy) or oxygen nightly. Participants receive the treatment expected to be most beneficial to them based on their baseline sleep study and OSA characteristics (OSA endotype).
  Interventions: Drug: ato-oxy; Drug: Oxygen

INTERVENTIONS:
Drug: ato-oxy — 0.5 mg/kg (max 40 mg) of atomoxetine and 5mg oxybutynin taken nightly.
  Other Names: atomoxetine and oxybutynin
Drug: Oxygen — Oxygen via nasal cannula used nightly
  Arms: Endotype Directed Treatment

SUMMARY:
Down syndrome is the most common genetic cause of intellectual disability. People with Down syndrome often have obstructive sleep apnea (OSA), a condition where people have difficulties with breathing while asleep. OSA can lead to poor sleep, worse quality of life, behavior problems and more difficulties with thinking ("cognitive impairment"). Current treatments for OSA in people with Down syndrome are not very effective or require surgery. The combination of 2 medications, atomoxetine and oxybutynin ("ato-oxy") is a promising treatment for OSA in people with Down syndrome, but ato-oxy does not work for everyone with Down syndrome. Similarly, oxygen is effective for OSA in some people, but does not work for everyone. This study will evaluate the use a precision medicine approach to increase the effectiveness of OSA treatment in people with Down syndrome. The study will compare two groups. In the first group, everyone will be treated with ato-oxy. In the second group, a precision medicine approach will be used to assign participants to either ato-oxy or oxygen therapy, based on the specific reasons they have OSA.

The research team will enroll 200 children (age 6-17 years old) and adults with Down syndrome and OSA from five sites across the country. Half of participants will randomly receive ato-oxy while the other will receive either oxygen or ato-oxy dependent upon which treatment would be expected to work better for them. The research team will measure OSA severity, quality of life, behavior and cognition at the start of the study and after 12 months of treatment for every participant. The study will also track any treatment side effects for each treatment group.

DETAILED DESCRIPTION:
Background and Significance: Obstructive sleep apnea (OSA) is one of the most common comorbidities present in individuals with Down syndrome. In children without Down syndrome, OSA has a prevalence of 2-5%2 whereas the prevalence of OSA in children with Down syndrome has been estimated at 50-79%. Similarly, OSA occurs in 12% of adults without Down syndrome, but occurs in 80-100% of adults with Down syndrome. In studies by our group and others, OSA has been associated with neurocognitive impairment and impaired health-related quality of life (HRQOL) in children and adults with Down syndrome. Cognition and HRQOL have been shown to improve with effective treatment of OSA in people with Down syndrome. However, current treatments for OSA have limited effectiveness in people with Down syndrome. Adenotonsillectomy has been shown to have limited efficacy, as 65-73% of children with Down syndrome have residual OSA after adenotonsillectomy. Similarly, positive airway pressure (PAP) effectiveness is limited by poor adherence. Hypoglossal nerve stimulation has emerged as a new treatment but is an invasive procedure that involves a surgically placed implant that many individuals may prefer to avoid. Additionally, surgical complications are more common in people with DS compared to people without Down syndrome. Use is also limited in younger children with significant growth remaining. Given this, there is a great need for effective alternative therapies. The combination of atomoxetine and oxybutynin (ato-oxy) is a promising alternative therapy but is not effective in all individuals with Down syndrome. Similarly, oxygen therapy is often considered as an alternative treatment for OSA but is not effective in all patients. Underlying physiologic patient characteristics (OSA endotype) have predicted treatment response for OSA with both ato-oxy and oxygen. OSA endotype-directed treatment appears to be a means to identify the right treatment for the right patient, which may have greater effectiveness compared to the same treatment for all individuals.

Study Aims: The goal of this study is to determine if a precision medicine approach, endotype-directed treatment, is more effective than a one-size fits all treatment approach (ato-oxy) for OSA in people with Down syndrome. Specific aims of the study include: Aim 1: To compare the effectiveness of ato-oxy therapy versus precision medicine (endotype-directed) treatment for OSA in people with Down syndrome over 12 months; Aim 2: To compare the effectiveness of ato-oxy versus precision medicine (endotype-directed) treatment approach for key patient-centered outcomes (PCOs), including health-related quality of life, behavior and cognition over 12 months; Aim #3: To compare the adverse effects of ato-oxy versus precision medicine (endotype-directed) treatment.

Study Description: This is a randomized clinical trial comparing ato-oxy versus endotype-directed treatment for OSA in children and adults with DS. We will enroll 200 participants with Down syndrome and OSA (100 children age 6-17 years, 100 adults age 18+ years). Participants will be recruited from five clinical sites from across the country as well as via outreach. Participants will be randomized 1:1 at an individual level to either ato-oxy or endotype-directed treatment, which would be either oxygen or ato-oxy dependent upon the individual's OSA endotype. The study primary outcome is obstructive apnea-hypopnea index, the primary measure of OSA severity. Secondary study outcomes include measures of HRQOL, behavior, cognition and adverse effects. Participants will receive treatment and be followed for a total of 12 months during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 years or older
2. Down syndrome diagnosis
3. Any gender or ethnicity
4. Adults without a legally authorized representative must have a caregiver/support person that can co-sign consent and complete study questionnaires.

Exclusion Criteria:

1. Currently using and adherent to PAP therapy (>4 hours per night for 70% of nights in the past 30 days based on device download or parent/caregiver report)
2. MAO inhibitor use
3. Urinary retention
4. Seizure disorder
5. Untreated or inadequately treated hypothyroidism
6. Significant traumatic brain injury
7. Not cleared to participate in the study by their cardiologist for individuals with congenital heart disease requiring follow up with cardiology at least once in the past year
8. History of current, untreated depression
9. History of liver disease (not including metabolic dysfunction-associated steatotic liver disease)
10. 3+ or greater tonsillar hypertrophy (for children only, no restriction for adults)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
obstructive apnea-hypopnea index (oAHI) | 12 months
  change in number of obstructive apneas and hypopneas per hour on polysomnography from baseline. Decreased oAHI indicates better outcome.

SECONDARY OUTCOMES:
Change in caregiver Pediatric Quality of Life (PedsQL) score from baseline | 12 months
  Change in caregiver reported quality of life as measured by PedsQL, higher scores indicate better outcome.
Change in Paired Associate Learning test total adjusted errors from baseline | 12 months
  Change in Paired Associate Learning test total errors (a measure of memory) from baseline. Fewer errors indicate better outcome

OTHER OUTCOMES:
Change in processing speed (Arizona Memory Assessment for Preschoolers and Special Populations [A-MAP] task) from baseline. | 12 months
  This is a computerized cognitive assessment. Faster processing speed indicates better outcome.
Change in total IQ (Kaufman Brief Intelligence Test 2) from baseline | 12 months
  Higher IQ indicates better outcome
Change in non-verbal IQ (Kaufman Brief Intelligence Test 2) from baseline | 12 months
  Higher IQ indicates better outcome
Change in verbal IQ (Kaufman Brief Intelligence Test 2) from baseline | 12 months
  Higher IQ indicates better outcome
Change in Arizona Memory Assessment for Preschoolers and Special Populations (A-MAP) verbal memory task from baseline | 12 months
  This is a computerized assessment of memory, higher scores indicate better outcome.
Change in expressive language from baseline | 12 months
  This will use the narrative generation task from the Expressive Language Sampling protocol. Narratives will be coded using an established scheme to capture detail generation, narrative length, and semantics. Longer narratives with more details and more correct semantics indicates better outcome.
Change in Caregiver Global Impression of Change from baseline | 12 months
  This is a single question on overall improvement. Higher reported improvement indicates better outcome.
Change in N1 sleep (%) from baseline | 12 months
Change in REM sleep (%) from baseline | 12 months
Change in N3 sleep (%) from baseline | 12 months
Change in arousal index (events/hr) from baseline | 12 months
Change in Vineland 3 adaptive behavior composite scale from baseline | 12 months
  Higher scores indicate better outcome.
Change in Conners-3 ADHD Index from baseline | 12 months
  Lower scores indicate better outcome
Change in self-reported Pediatric Quality of Life Inventory (PedsQL) total score | 12 months
  Change in self-reported quality of life as measured by PedsQL
Change in caregiver-reported Pediatric Quality of Life Inventory (PedsQL) family impact | 12 months
Hypoxic burden | 12 months
  Desaturation area under curve × event frequency, lower burden indicates better outcome.
Ventilatory burden | 12 months
  The proportion of breaths during sleep with less than 50% of their normal amplitude
Supine obstructive apnea-hypopnea index (oAHI) | 12 months
  obstructive apnea-hypopnea index while sleeping supine. Lower oAHI indicates better outcome.
non-supine obstructive apnea-hypopnea index (oAHI) | 12 months
  obstructive apnea-hypopnea index while sleeping in any position other than supine. Lower oAHI indicates better outcome.
total Apnea Hypopnea Index (AHI) | 12 months
  Lower AHI indicates better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Combs, MD, Principal Investigator — University of Arizona
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - University of Miami, Miami, Florida
  - Advocate Medical Group Adult Down Syndrome Center, Park Ridge, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available.

REFERENCES:
- [Background] Combs D, Edgin J, Hsu CH, Bottrill K, Van Vorce H, Gerken B, Matloff D, La Rue S, Parthasarathy S. The combination of atomoxetine and oxybutynin for the treatment of obstructive sleep apnea in children with Down syndrome. J Clin Sleep Med. 2023 Dec 1;19(12):2065-2073. doi: 10.5664/jcsm.10764. PMID 37555595